CLINICAL TRIAL: NCT01268839
Title: A Phase I, Open-label Trial to Explore the Pharmacokinetics, Safety and Tolerability of TMC278 25 mg Once Daily Following a 2-week Period Receiving Efavirenz, in Healthy Male and Female Subjects
Brief Title: A Phase I, Open-label Trial to Explore the Pharmacokinetics, Safety and Tolerability of TMC278 (Rilpivirine) 25 mg Once Daily Following a 2-week Period Receiving Efavirenz, in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec, Inc (Industry)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR016984; TMC278HIV1001
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: HIV
Keywords: TMC278, rilpivirine, efavirenz, healthy volunteer
MeSH Terms: interventions — Rilpivirine; efavirenz

ARMS (1):
- 001 (Experimental): Efavirenz 600mg tablet once daily for 14 days,TMC278 25mg tablet once daily for 14 days,TMC278 25mg tablet once daily for 28 days
  Interventions: Drug: TMC278; Drug: Efavirenz

INTERVENTIONS:
Drug: TMC278 — 25mg tablet once daily for 28 days
Drug: TMC278 — 25mg tablet once daily for 14 days
Drug: Efavirenz — 600mg tablet once daily for 14 days

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of TMC278 (rilpivirine) 25 mg once daily following a preceding 2-week treatment period with efavirenz 600 mg once daily in healthy volunteers

DETAILED DESCRIPTION:
This is a Phase I, open-label (all people involved know the identity of the intervention), single center trial in healthy HIV negative volunteers to investigate the pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body, the rate at which a drug action begins, the duration of the effect, the chemical changes of the substance in the body, and the effects and routes of excretion of the metabolites) of the drug of rilpivirine (TMC278) 25 mg once daily (q.d.). An approximate total of 20 volunteers will be enrolled in this trial. All volunteers will receive 3 different treatments; o Treatment A: TMC278 25 mg q.d. administered for 14 days.; o Treatment B: efavirenz (EFV) 600 mg q.d. administered for 14 days.; o Treatment C: TMC278 25 mg q.d. administered for 28 days (4 weeks).; All volunteers will start with Treatment A followed by Treatment B. Treatments A and B will be separated by a washout period of at least 14 days but no more than 21 days. At the end of Treatment B, volunteers will continue with Treatment C. There will be no washout period between Treatments B and C.; Full pharmacokinetic profiles of TMC278 will be determined up to 24 hours postdose on Days 1 and 14 of Treatment A (references), Day 1 (immediately after cessation of EFV intake) of Treatment C (test), and on Days 14, 21, and 28 (2, 3, and 4 weeks after cessation of EFV intake, respectively) of Treatment C. Trough (C0h) samples for determination of TMC278 plasma; concentrations will be collected regularly in between. Blood samples for determination of EFV plasma concentrations will be collected at regular time points during Treatment B and during Treatment C after cessation of EFV intake.; Serum samples for potential future testing of ex vivo antiviral activity will be collected and stored.; A pharmacogenomic blood sample for potential future CYP2B6 genotyping will be collected and stored from subjects who consent separately to the pharmacogenomic component of the trial.; Safety and tolerability will be evaluated throughout the trial. Rilpivirine (TMC278) 25mg once daily for 14 days, No Treatment 14-21 days, Efavirenz 600mg once daily for 14 days, TMC278 25mg once daily for 28 days

ELIGIBILITY:
Inclusion Criteria:

* Non-vasectomized heterosexually active male volunteers with female partner of childbearing potential must be using a highly effective method of birth control (i.e., male condom with either female intrauterine device, diaphragm, cervical cap or hormonal based contraceptives) and must agree to use these birth control methods during the trial and until 30 days after the end of the trial
* Able to comply with all protocol requirements
* Normal resting ECG at screening including
* Volunteers must have signed an Informed Consent Form (ICF) voluntarily before the first trial-related activity indicating that they understand the purpose of and procedures required for the trial and are willing to participate in the trial
* To participate in the optional pharmacogenomic component of this trial, volunteers must have signed the ICF for pharmacogenomic research indicating willingness to participate in the pharmacogenomic component of the trial. Refusal to give consent for this component does not exclude a volunteers from participation in the clinical trial
* Healthy on the basis of a medical evaluation that confirms the absence of any clinically relevant abnormality and includes a physical examination (including skin examination), medical history, vital signs, the results of blood biochemistry and hematology tests and a urinalysis carried out at screening.

Exclusion Criteria:

* A positive HIV-1 or -2 test at trial screening
* Females of childbearing potential
* Hepatitis A infection (confirmed by hepatitis A antibody IgM), hepatitis B infection (confirmed by hepatitis B surface antigen), or hepatitis C infection (confirmed by hepatitis C virus antibody) diagnosed at trial screening
* Currently active clinically significant disease (e.g., pancreatitis, cardiac dysfunction) or findings during screening of medical history, laboratory or physical examination that in the investigator's opinion would compromise subject safety or the outcome of the trial
* Current or recent (within 3 months prior to the first administration of trial medication) gastrointestinal disease
* Any history of significant skin disease such as but not limited to rash or eruptions, drug allergies, food allergy, dermatitis, eczema, psoriasis, or urticaria
* A positive alcohol test or urine drug test at study screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of TMC278 25 mg once daily (q.d.) following a preceding 2-week treatment period with EFV 600 mg q.d., in healthy volunteers | 70-77 days

SECONDARY OUTCOMES:
To evaluate the EFV inducing effect on TMC278 metabolism after EFV intake cessation, through comparison of TMC278 plasma concentrations with and without preceding EFV intake | 70-77 days
To evaluate EFV plasma concentrations over time after cessation of EFV intake | 70-77 days
To assess the safety (including vital signs and electrocardiogram [ECG] measurements, laboratory assessments, and incidence of overall AEs and tolerability) of TMC278 at a dose of 25 mg q.d administered alone and after switching from EFV over a period of | 70-77 days

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec, Inc. Clinical Trial, Study Director — Tibotec, Inc